CLINICAL TRIAL: NCT03697915
Title: Implementing Lift System to Physical Therapy Program for Early Mobilization in Immobilised Patients: A Randomised Controlled Trial
Brief Title: Implementing Lift System for Early Mobilization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, TOMRIS DUYMAZ, Asst. Prof. Ph.D., Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-40016-46
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Inpatient Facililty Diagnoses
Keywords: Lift system; Early mobilization; Immobilization

STUDY DESIGN:
Intervention Model Description: Thirty hospitalized patients who were immobile more than 1 week were randomised into two groups. Each group had received 15 sessions of physical therapy (ROM exercises and electrotherapy) regularly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group, in which a physical therapy programme supplemented by the James lift system was applied
  Interventions: Device: Experimental
- Control (Placebo Comparator): Control group, in which a conventional physical therapy programme was applied.
  Interventions: Device: Experimental

INTERVENTIONS:
Device: Experimental — Conventional physical therapy was administered to the control group and was aimed at achieving sitting balance in the first phase; once sitting balance could be achieved, we aimed at achieving standing balance in the second phase. Once standing balance was also achieved, supported and unsupported ambulation was commenced in the final phase.
  Other Names: Control

SUMMARY:
Objective:Immobilization causes various physiological and biomechanical problems during inpatient treatments.Physical therapy is applied to achieve early mobilization and avoid complication of immobilization.

Aim:The aim of this study is to assess the contribution of using lift system to physical therapy program of immobilized patients.

Design:A randomised controlled trial. Patients:Thirty hospitalized patients who were immobile more than 1 week were randomised into two groups.

Interventions: Each group had received 15 sessions of physical therapy (ROM exercises and electrotherapy) regularly.Patients allocated to the add-on lift system were held in upright position with James lift® system during each physical therapy(PT).Patients allocated to PT program only were upgraded to a therapeutic goal of stability during standing phase as the patient's muscular strength improved.

DETAILED DESCRIPTION:
In this study, 30 patients aged 50-75 years who were immobilised for >1 week and were conscious but did not have sitting balance were evaluated. Before this study was initiated, approval was obtained from the XXX University Ethics Committee (number 2018-40016-46, dated 24/04/2018). The inclusion criteria for the study included having undergone surgical procedures leading to immobilisation or having a disease affecting the musculoskeletal system, being conscious and not having sitting balance. The exclusion criteria included co-operation, orientation and cognitive impairment.

Patients were divided into two groups: control group, in which a conventional physical therapy programme was applied, and experimental group, in which a physical therapy programme supplemented by the James lift system was applied. Randomisation was performed according to the hospitalisation order of the patients.

Conventional physical therapy was administered to the control group and was aimed at achieving sitting balance in the first phase; once sitting balance could be achieved, we aimed at achieving standing balance in the second phase. Once standing balance was also achieved, supported and unsupported ambulation was commenced in the final phase.

In addition to the conventional treatment programme in the experimental group, orthostatic blood pressure was checked at the early stage before the patients gained sitting balance. Once the patients gained standing balance using the lift, they were administered walking training.

Conventional physical therapy was administered to both the groups and included passive and active assisted joint range of motion exercises, sitting balance, standing balance, electrotherapy (20 min of electrical stimulation on bilateral quadriceps and muscles) and ambulatory training.

Pre- and post-treatment evaluations included age, height, weight, duration of hospital stay and day of initial mobilisation. Clinical and Rivermead mobility indices were used as the primary outcome. The Barthel index, which assesses daily living activities, and hospitalisation period were evaluated as secondary outcomes.

The James 150 lift system is a hydraulic system made of steel pipes with a carrying capacity of 150 kg and is designed to keep the patients in an upright position. It is a hydraulic transport system with a short installation time, including an electric lift arm, 24-Volt motor, wired remote control, emergency button, mechanical emergency lowering, extensible undercarriage pedal, swivel castors and rear-wheel brakes. When a patient is required to be switched to the upright position, he/she is supported by Velcro sheaths in the thoracolumbar area, knees are locked with knee supports, feet are switched to the dorsiflex position using the foot pedal and the patient is brought to the upright position. During this time, the patient grips the lift handles with his/her hands for support. The patient is protected against falling during the lifting process by the brake-lock system.

The Rivermead mobility index reflects basic mobility activities. The questionnaire consists of 15 questions, of which 14 are self-reported items and one is a direct observation item. "Yes" answers are given 1 point. The index is scored between 0 and 15 points, where 15 indicate normal mobility, whereas ≤14 indicate impaired mobility.

The clinical mobility scale evaluates the level of mobility and is scored between 0 and 3 points. It includes the following items: upright posture, walking, gait, sitting, stair climbing, hand-held appliances and wheelchair and time usage. It is scored between 0 and 24 points, and higher scores indicate increased mobility.

The Barthel index scores daily life activities. The total score can range between 0 and 100 points, with each question score ranging from 0.5 to 10 points. The sub-topics covered include feeding, bathing, grooming, dressing, bowel care, bladder care, toilet use, transfer (bed to chair and back), mobility (on levelled surfaces) and stair climbing. Higher scores indicate improved independence of the patient.

ELIGIBILITY:
Inclusion Criteria:

* undergone surgical procedures leading to immobilisation
* having a disease affecting the musculoskeletal system
* being conscious and not having sitting balance.

Exclusion Criteria:

* co-operation, orientation
* cognitive impairment.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-06-02 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-10-08 (Estimated)

PRIMARY OUTCOMES:
Mobility index | 1 minute
  The Rivermead mobility index reflects basic mobility activities. The questionnaire consists of 15 questions, of which 14 are self-reported items and one is a direct observation item. "Yes" answers are given 1 point. The index is scored between 0 and 15 points, where 15 indicate normal mobility, whereas ≤14 indicate impaired mobility

SECONDARY OUTCOMES:
Daily life activities | 3 minutes
  The Barthel index scores daily life activities. The total score can range between 0 and 100 points, with each question score ranging from 0.5 to 10 points. The sub-topics covered include feeding, bathing, grooming, dressing, bowel care, bladder care, toilet use, transfer (bed to chair and back), mobility (on levelled surfaces) and stair climbing. Higher scores indicate improved independence of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Tomri̇s Duymaz, Principal Investigator — Istanbul Bilgi University
Locations (1):
- Tomri̇s Duymaz, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided